CLINICAL TRIAL: NCT03520634
Title: PD-L1 PET Imaging in Patients With an Inoperable Melanoma With Brain Metastasis and Eligible for Treatment With Nivolumab.
Brief Title: PD-L1 PET Imaging in Melanoma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 31052016
Record Dates: First submitted 2016-05-31; First posted 2018-05-11 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2021-04

CONDITIONS: Melanoma
Keywords: Melanoma; PD-L1; Brain metastases; PET imaging
MeSH Terms: conditions — Melanoma; Brain Neoplasms | interventions — BMS-986192

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-L1 PET imaging in melanoma patients (Experimental): The main intervention of this study is a [18F]PD-L1 PET scan. In both phase one and phase two a scan sequence will be performed both at baseline and 6 weeks after initiation of nivolumab treatment. The PET scans will be combined with either a low dose or diagnostic CT scan of chest, abdomen and pelvis and a MRI of the brain. In phase two, a biopsy of at least one accessible lesion will be performed to analyze PD-L1 expression using immunohistochemical staining after each PET scan.
  Interventions: Other: PD-L1 PET imaging

INTERVENTIONS:
Other: PD-L1 PET imaging — PD-L1 PET imaging
  Other Names: [18F]BMS-986192

SUMMARY:
This is a feasibility study for the use of [18F]PD-L1 as a PET tracer that will be conducted in a single center. The study consists of two phases. The aim of phase one is to provide pharmacokinetic information on the tracer and to determine the optimal time point for imaging. In the second phase the main study objective will be assessed.

DETAILED DESCRIPTION:
This is a single center feasibility study for the application of [18F]PD-L1 PET in patients with metastatic melanoma and NSCLC treated with anti-PD-1 therapy. The study will consist of a pharmacokinetics phase (phase one) and tracer validation phase (phase two). Phase one will be performed in a maximum of 5 patients. A [18F]PD-L1 PET scan will be performed at baseline and six weeks after treatment initiation. Upon finishing phase one, the optimal time for tracer injection will bedetermined prior to the start of phase two. In phase two a [18F]PD-L1 PET-CT scan will be performed in 10 patients at baseline and six weeks after treatment initiation. Also, when it is feasible a biopsy will be taken from at least one accessible tumor location after the PET-scan at baseline and the PET-scan after six weeks of therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must sign informed consent prior to inclusion in this trial.
2. Subjects must be ≥18 years of age and competent to give informed consent.
3. Subjects must be diagnosed with histologically confirmed stage IV melanoma.
4. At least one radiologic new lesion in the brain by MRI, which should be measurable by RANO-BM criteria (longest diameter ≥ 10 mm and perpendicular diameter ≥ 5 mm). Lesions with prior local treatment (i.e., SRT or surgical resection) can be considered measurable if there has been demonstrated progression since the time of local treatment. Leptomeningeal involvement is allowed, but cannot be used as target lesion.
5. At least one easy accessible metastatic melanoma lesion of which a biopsy can be taken.
6. Subjects must be treatment-naive to nivolumab. (also as adjuvant treatment)
7. Subjects must score at least 1 or higher on the Eastern Cooperative Oncology Group (ECOG) Performance Status.(21)
8. Subjects must have adequate organ function as defined by the following laboratory values (determined within 28 days prior to randomization/registration):

   * White blood cells (WBC) ≥ 2000 /μL
   * Absolute neutrophil count (ANC) ≥ 1500 /μL
   * Platelets ≥ 100 x103 /μL
   * Hemoglobin ≥ 9 g/dL or ≥ 5.6 mmol/L
   * Serum creatinine ≤ 1.5 times upper limit of normal (ULN) or creatinine clearance > 40 ml/min (using the Cockcroft-Gault formula)
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 times ULN
   * Bilirubin ≤ 1.5 times ULN (Except patients with the Gilbert Syndrome, for whom a maximum of ≤ 3.0 mg/dL is acceptable)
9. Women of childbearing potential (WOCBP) should have a negative urine or serum pregnancy test within 7 days prior to receiving the first administration of nivolumab. Women with non-childbearing potential may be included if they are either surgically sterile or have been postmenopausal for ≥ 1 year.
10. WOCBP and men who are sexually active with WOCBP must agree to use appropriate method(s) of contraception. (see section 5.2)

Exclusion Criteria:

1. Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2 antibody, or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways, except anti-CTLA4 antibody.
2. Subjects who have not recovered to Common Terminology Criteria for Adverse Events (CTCAE) v4.0 Grade 1 or better from the adverse events due to previous cancer therapy.
3. Evidence for an active, known or suspected autoimmune disease. Subjects diagnosed with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
4. Treatment with corticosteroids in an increasing dosage in the 7 days prior to the first administration of nivolumab. (A stable or decreasing dosage of ≤ 4 mg dexamethasone or equivalent is allowed. In addition, inhaled or topical steroids and adrenal replacement doses are permitted in the absence of active autoimmune disease.)
5. Previous malignancies (except non-melanoma skin cancers, in situ bladder cancer, gastric or colon cancers, cervical cancers/dysplasia or breast carcinoma in situ) unless a complete remission was achieved at least 1 years prior to study entry and no additional therapy is required or anticipated to be required during the study period.
6. A severe hypersensitivity reaction to prior treatment with a monoclonal antibody, or known hypersensitivity to study drugs components.
7. A positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection.
8. Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
9. Any serious or uncontrolled medical disorder or active infection that, in the opinion of the investigator, may increase the risk associated with study participation, study drug administration, or would impair the ability of the patients to receive protocol therapy.
10. A known psychiatric or substance abuse disorder that could interfere with cancer therapy.
11. Women of childbearing potential with a positive serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of nivolumab.
12. Breastfeeding women.
13. Inability to comply with other requirements of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2021-04-12 (Actual)

PRIMARY OUTCOMES:
Determine the optimal dose of tracer and timing of imaging for [18F]PD-L1 tracer imaging of inoperable melanoma. | 1 year
  By the performing dynamic PET scans.
Assess the association of PD-L1 expression as measured by PD-L1 tracer uptake on PET and PD-L1 expression as measured by immunohistochemical (IHC) staining for PD-L1 of corresponding tumor lesions. | 1 year
  By the performing Full body PET scans.

SECONDARY OUTCOMES:
Characterize between-subject and within-subject variability in accumulation of the [18F]PD-L1 tracer in melanoma metastases. | 1 year
  By the quantification of Full body PET scans.
Correlate response to anti-PD1 treatment with differences in tumor PD-L1 and PD1 expression between baseline and after 6 weeks of treatment. | 1 year
  As quantified by PET and IHC analysis.

CONTACTS AND LOCATIONS:
Overall Officials: G.A. P Hospers, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- UMCG, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-20): https://cdn.clinicaltrials.gov/large-docs/34/NCT03520634/Prot_SAP_000.pdf